CLINICAL TRIAL: NCT06005220
Title: A Randomised, Double Blind Placebo-controlled Trial Evaluating the Medical Food Synbiotic SBD121, Versus Placebo for the Clinical Dietary Management of Early Rheumatoid Arthritis.
Brief Title: SBD121, a Synbiotic Medical Food for RA Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solarea Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SOL-SYNBIOTIC-2023
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBD121 Medical Food (Active Comparator): Two capsules administered twice daily with food
  Interventions: Other: SBD121
- Placebo (Placebo Comparator): Two capsules administered twice daily with food
  Interventions: Other: Placebo

INTERVENTIONS:
Other: SBD121 — Medical Food
  Arms: SBD121 Medical Food
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this randomised, double-blind, placebo controlled clinical food trial is to determine if the medical food SBD121 Synbiotic (prebiotic and probiotic) will aid in the dietary management of symptoms of early rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to the performance of any study-specific procedure and willing to comply with the protocol and report on compliance and side effects during study period.
2. Male or female aged 18 - 75 years inclusive at the time of consent.
3. The participant must have newly diagnosed RA, not exceeding 1-year from diagnosis
4. The participant must have been taking methotrexate (MTX) for treatment of RA for ≤ 75 days before baseline, or will be commencing MTX at the same time as baseline (within range 15 to 25 mg inclusive, recommended target dose of 20mg).
5. The participant must have active RA meeting classification criteria according to the 2010 ACR/EULAR guidelines with a score equal to or greater than 6/10 at screening (11). (Seropositivity is not required).
6. The participant must be available throughout entire study period, willing and able to attend all scheduled visits and in the opinion of the Investigator be able to understand and comply with planned study procedures.
7. Body Mass Index (BMI) between 18.5 and 40 kg/m2
8. Normal cardiovascular parameters (systolic blood pressure ≤ 150 mm Hg, diastolic blood pressure ≤ 90 mm Hg). One re-test is permitted.
9. Women of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test pre-first administration, on Day 1, and must agree to remain sexually abstinent, or use medically effective contraception (refer to Appendix 11.1), or have a partner who is sterile or same-sex, from Screening until end of study. Males must not be planning to father children or donate sperm for the duration of the study.

Exclusion Criteria:

1. Participant is currently taking any probiotic or prebiotic supplements, or has taken them in the past 7 days, or is unwilling to avoid taking probiotic/prebiotic supplements for the duration of the study.
2. Participant has any known or suspected allergies to probiotics or prebiotics.
3. Participant has taken oral or parenteral antibiotics within 21 days of screening, requires antibiotics pre-first dose, or is likely to require antibiotics during the study period.
4. Participant has undergone major surgery within last 3-months before screening or planned during the study period
5. Participant is a current or past smoker and/or user of nicotine replacement therapies (including vaping), that in the documented opinion of the Investigator, may adversely affect participation in the study, safety, and/or study outcomes.
6. Participant has a past or current history of drug and/or alcohol abuse at the time of enrolment (the use of illegal drugs or the use of prescription or over-the-counter drugs or alcohol for purposes other than those for which they are meant to be used, or in excessive amounts).
7. Participant has a known history of any of the following (according to Investigator judgement and/or participant report):

   1. Gastric or intestinal dysmotility, slowed transit time, pancreatitis, or inflammatory bowel disease
   2. Known Hepatitis B or Hepatitis C infection, cirrhosis or chronic liver disease
   3. Underlying structural heart disease or previous history of endocarditis or valve replacement
   4. Rheumatic disease other than rheumatoid arthritis, including but not limited to psoriasis, spondyloarthritis, systemic lupus erythematosus, multiple sclerosis
   5. Immunosuppressed, including: known HIV positive; solid organ or stem cell transplant recipient; taking any oral or parenteral immunosuppressive therapy; neutrophil count <500/mm3; or anticipated drop in the neutrophil count to <500/mm3
   6. Any malignancy, with the exception of non-melanoma skin cancers, or other cancer more than 5-years ago
   7. Active tuberculosis (TB) within 3-months prior to Screening
   8. Any infection requiring hospitalisation, or as otherwise judged clinically significant, within 3-months prior to Screening
8. Presence of any of the following active conditions at Screening, or within 72 hours of the first administration of study test article:

   1. Clinically significant abnormal vital signs or physical examination abnormalities (other than those related to RA, such as joint swelling)
   2. Febrile illness (temp. > 37.5 degrees Celsius), or one or more episodes of diarrhoea within 72 hours of the first dose of study test article
   3. Acute abdomen, colitis, or active GI disease
   4. Septicaemia or bacteraemia
   5. Uncontrolled diabetes mellitus, based on medical history and in response to query 'is your diabetes under control?'.
9. Current treatment with any Disease Modifying Arthritis Drug (DMARD) other than methotrexate including but not limited to, hydroxychloroquine, sulfasalazine, and minocycline leflunomide, gold compounds, azathioprine, or cyclosporine will be exclusionary if used within 30 days prior to randomisation.
10. Current or past treatment with any biologic agent including but not limited to tumor necrosis factor (TNF) inhibitors: etanercept, infliximab, adalimumab; interleukin 1 (IL-1) inhibitors: anakinra; lymphocyte directed: abatacept, rituximab; Janus kinase (JAK) inhibitors: tofacitinib; interleukin 17 (IL-17) inhibitors; Interleukin 23 (IL-23) inhibitors.
11. Corticosteroid use from 30 days prior to randomisation until final assessment visit will be exclusionary, with the following exceptions:

    1. Oral corticosteroids in low doses (≤ 10 mg/d prednisone or equivalent) will be allowed if stable for 1-month prior to randomisation. Reduction of dose or use of oral corticosteroids is permissible throughout the study.
    2. Topical, inhaled, or intranasal steroids are permitted
    3. Past use of oral or parenteral (> 10 mg/d prednisone or equivalent) corticosteroids is allowed if not used within 1-month prior to randomisation.
12. Women only - pregnant, planning on becoming pregnant during the trial, breastfeeding, positive urine pregnancy test during Screening or within 24 hours of first administration of study test article.
13. Any of the following abnormal findings on Screening or Baseline laboratory tests (one re-test per timepoint permitted):

    1. White blood cells (WBCs) < lower limit of normal (LLN) or > upper limit of normal (ULN). If WBC is documented within normal range prior to commencing steroids and is deemed by the Investigator as elevated at screening due to recent addition of these drugs and not related to any other comorbidities, then may be suitable to proceed.
    2. Neutrophils < 1500/µl (1.5 x109/L)
    3. Platelets < 100 x 10³/µl (100 x 109/L)
    4. Haemoglobin < 9.0 g/dl (90 g/L)
    5. Serum Creatinine > 1.5 x ULN
    6. Glomerular filtration rate (GFR) of < or = 40 mL/minute
    7. Aspartate aminotransferase (AST) > 3 x ULN
    8. Alanine aminotransferase (ALT) > 3 x ULN
    9. Total Bilirubin > 1.5 x ULN
14. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer participating in the study or would make it unlikely the volunteer could complete the study
15. If the participant has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 20 (ACR-20) | 16 Weeks
  Evaluate the dietary management of arthritis by the number and percentage of participants achieving American College of Rheumatology 20 (ACR20) response (ie, greater to or equal to 20% improvement in the ACR composite score, a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, arthritis activity, and physical function; physician's assessment of arthritis activity; and CRP) at Week 16

SECONDARY OUTCOMES:
Safety by Adverse Events | 16-weeks
  Number and percentage of participants experiencing adverse events (AEs) and serious adverse events (SAEs)
Tolerability by GITQ | 16-weeks
  Frequency and severity of GI symptoms (e.g., gas, abdominal pain, bloating) as assessed by the Gastrointestinal Tolerability Questionnaire (GITQ) score at each timepoint compared to placebo.
American College of Rheumatology 20 (ACR-20) | 8 weeks
  Evaluate the dietary management of arthritis by the number and percentage of participants achieving American College of Rheumatology 20 (ACR20) response (ie, greater to or equal to 20% improvement in the ACR composite score, a measure of RA symptoms including: joint swelling and tenderness; patient's assessment of pain, arthritis activity, and physical function; physician's assessment of arthritis activity; and CRP) at Week 8
American College of Rheumatology 50 (ACR-50) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the number and percentage of participants achieving ACR50 response in the ACR composite score at Week 8, and Week 16
American College of Rheumatology 70 (ACR-70) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the number and percentage of participants achieving ACR70 response in the ACR composite score at Week 8, and Week 16
Disease Activity Score 28 - Eosinophil Sedimentation Rate (DAS28 - ESR) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the percentage change from baseline value in the Activity Score-28 (DAS-28) with ESR (DAS-28-ESR), and the individual components that make up the DAS-28-ESR [Tender Joint Count (TJC), Swollen Joint Count (SJC), and Patients Global Assessment of Activity, plus Erythrocyte Sedimentation Rate (ESR)], at 8 and 16 weeks
Disease Activity Score 28 - C-Reactive Protein (DAS28 - CRP) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the percentage change from baseline value in the DAS-28 with CRP score and the individual components that make up the DAS-28 CRP Score [Tender Joint Count (TJC), Swollen Joint Count (SJC), and Patients Global Assessment of Activity, plus C-Reactive Protein (CRP)], at 8 and 16 weeks
Disease Activity Score 28 - Eosinophil Sedimentation Rate - Low Disease Activity (DAS28 - ESR - LDA) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the percentage of participants who achieve DAS-28-ESR Low Activity defined as DAS-28-ESR Score < 3.2, at 8 and 16 weeks
Disease Activity Score 28 - C-Reactive Protein - Low Disease Activity (DAS28 - CRP LDA) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the percentage of participants who achieve DAS-28-CRP Low Activity, defined as DAS-28-CRP Score < 3.2, at 8 and 16 weeks
Disease Activity Score 28 - Eosinophil Sedimentation Rate - Remission (DAS28 - ESR Remission) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the percentage of participants who achieve DAS-28-ESR Remission defined as DAS-28-ESR Score < 2.6, at 8 and 16 weeks
Disease Activity Score 28 - C-Reactive Protein - Remission (DAS28 - CRP Remission) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the percentage of participants who achieve DAS-28-CRP Remission, defined as DAS-28-CRP Score < 2.6, at 8 and 16 weeks
C-Reactive Protein (CRP) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the improvement in CRP from baseline
Eosinophil Sedimentation Rate (ESR) | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the improvement in ESR from baseline
Zonulin | 8-weeks, 16-weeks
  Evaluate improvement in gastrointestinal permeability by improvement in Zonulin from baseline
Reduce or discontinue use of oral corticosteroids | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the number and percentage of participants able to reduce dose or discontinue use of oral corticosteroids, at 8 and 16 weeks
Reduce or discontinue use of oral NSAIDs | 8-weeks, 16-weeks
  Evaluate the dietary management of arthritis by the number and percentage of participants able to reduce dose or discontinue use of oral NSAIDs, at 8 and 16 weeks

OTHER OUTCOMES:
Microbiome functional composition by shotgun metagenomics | 16-weeks
  Change in the functional gut microbiota composition in stool samples from baseline and correlation with primary and secondary efficacy outcomes, at 16 weeks
Microbiome taxonomic composition by shotgun metagenomics | 16-weeks
  Change in the taxonomic gut microbiota composition in stool samples from baseline and correlation with primary and secondary efficacy outcomes, at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Stanley, Study Director — Southern Star Research
Locations (22):
- Australia (12):
  - Paratus Clinical Canberra, Canberra, Australian Capital Territory
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Genesis Research Services, Newcastle, New South Wales
  - BJC Health, Parramatta, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St. Vincents Hospital Melbourne, Melbourne, Victoria
  - Western Health, St Albans, Victoria
  - Linear Clinical Trials, Nedlands, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- Bulgaria (5):
  - Diagnostic Consultative Center 1 - Lom EOOD, Lom
  - Medical Center - Teodora EOOD, Rousse
  - MHAT Lyulin EAD, Department of Rheumatology, Sofia
  - Diagnostic Consultative Center XIV - Sofia EOOD, Sofia
  - Medical Center Tera Medico EOOD, Vrasta
- Moldova (2):
  - RTL SM SRL/ IMSP Institutul de Cardiologie, Chisinau
  - Spitalul Clinic Republican Timofei Mosneaga, Chisinau
- New Zealand (3):
  - Aotearoa Clinical Trials, Auckland
  - Optimal Clinical Trials, Auckland
  - Southern Clinical Trials, Nelson

IPD SHARING:
Plan to Share IPD: No